CLINICAL TRIAL: NCT03703063
Title: Alternating Neoadjuvant Gemcitabine-Nab-Paclitaxel and Nanoliposomal Irinotecan (Nal-IRI) With 5-Fluorouracil and Folinic Acid (Leucovorin) Regimens in Resectable and Borderline Resectable Pancreatic Cancer
Brief Title: Alternative Neoadjuvant Chemotherapy in Resectable and Borderline Resectable Pancreatic Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benaroya Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRP17118
Record Dates: First submitted 2018-10-08; First posted 2018-10-11 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic cancer; nal-IRI; NAPOLI
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Taxes; Albumin-Bound Paclitaxel; irinotecan sucrosofate; Leucovorin; Fluorouracil

STUDY DESIGN:
Intervention Model Description: Resectable patients And Borderline resectable patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Resectable patients (Experimental): Gemcitabine and Nab-Paclitaxel Participants received albumin-bound paclitaxel 125 mg/m^2 followed by gemcitabine 1000 mg/m^2 by intravenous infusion (IV) on Days 1, 8 and 15 of each 28 day cycle. Followed by nal-IRI (ONIVYDE®) 70 mg/m^2 followed by leucovorin 400 mg/m^2 followed by 5FU 2400 mg/m^2 on days 1, 15 of the 28 day cycle.
  Interventions: Drug: Gemcitabine; Drug: nab paclitaxel; Drug: Onivyde; Drug: Leucovorin; Drug: 5-fu
- Borderline resectable patients (Experimental): Gemcitabine and Nab-Paclitaxel Participants received albumin-bound paclitaxel 125 mg/m^2 followed by gemcitabine 1000 mg/m^2 by intravenous infusion (IV) on Days 1, 8 and 15 of each 28 day cycle. Followed by nal-IRI (ONIVYDE®) 70 mg/m^2 followed by leucovorin 400 mg/m^2 followed by 5FU 2400 mg/m^2 on days 1, 15 of the 28 day cycle.
  Interventions: Drug: Gemcitabine; Drug: nab paclitaxel; Drug: Onivyde; Drug: Leucovorin; Drug: 5-fu

INTERVENTIONS:
Drug: Gemcitabine — Administered by intravenous infusion over 30 minutes.
  Other Names: Gemzar
Drug: nab paclitaxel — Administered by intravenous infusion over 30-40 minutes.
  Other Names: Abraxane
Drug: Onivyde — Administered by intravenous infusion over 90 minutes.
Drug: Leucovorin — Administered by intravenous infusion over 30 minutes.
Drug: 5-fu — Administered by intravenous infusion over 46 hours.

SUMMARY:
Using alternative neoadjuvant gemcitabine-nab-paclitaxel and nal-IRI with 5-Fluorouracil (5FU) and folinic acid (Leucovorin) regimens of localized cancer, we hope to ensure exposure of the cancer to a broader array of potentially active agents. Also, potentially improves patient tolerance and minimizes significant drug toxicity that could impair delivery of all treatment elements. Furthermore, it may enable prediction of superior to inferior treatment outcomes at an earlier point in the disease progress.

DETAILED DESCRIPTION:
This research study is a Phase Ib clinical trial. It will assess the Safety, tolerability, and feasibility of gemcitabine-nab paclitaxel alternating with nal-IRI/5FU/leucovorin (NAPOLI) in de novo resectable and borderline resectable pancreatic cancer.

Subjects must have a newly diagnosed resectable or borderline resectable pancreatic ductal cancer and meet all inclusion/exclusion criteria.

Treatment consists of 4 week treatment cycles. Nab-paclitaxel and gemcitabine will be administered on days 1,8, and 15 with NAPOLI will be administered on days 1 and 15.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven resectable or borderline resectable pancreatic cancer per current NCCN criteria (http://www.nccn.org/professionals/physician_gls/f_guidelines.asp).
2. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0/1.
3. Adequate bone marrow reserves as evidenced by:

   * absolute neutrophil count (ANC) ≥1,500 cells/μl without the use of hematopoietic growth factors; and
   * Platelet count ≥100,000 cells/μl; and
   * Hemoglobin ≥9 g/dL (blood transfusions are permitted for patients with hemoglobin levels below 9 g/dL).
4. Adequate hepatic function as evidenced by:

   * Serum total bilirubin within normal range for the institution (biliary drainage is allowed for biliary obstruction); and
   * aspartate aminotransferase (AST) and alanine aminotransferase (ALT)

     * 2.5 x upper limit of normal (ULN) (≤5 x ULN is acceptable if liver metastases are present).
5. Adequate renal function as evidenced by a serum creatinine ≤1.5 x ULN.
6. At least 18 years of age.
7. Women of child-bearing potential (defined as a sexually mature woman who (1) has not undergone hysterectomy [the surgical removal of the uterus] or bilateral oophorectomy [the surgical removal of both ovaries] or (2) has not been naturally postmenopausal for at least 24 consecutive months [i.e., has had menses at any time during the preceding 24 consecutive months]) must: Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis), or agree to use, and be able to comply with, effective contraception without interruption for 28 days prior to starting study medications (including dose interruptions) and for 3 months after last dose of study medication and Have a negative pregnancy test result at screening and agree to ongoing pregnancy testing at the Investigator's discretion during the course of the study. This applies even if the subject practices true abstinence from heterosexual contact.
8. Male subjects must practice true abstinence or agree to use a condom during sexual contact with a female of childbearing potential or a pregnant female while on treatment (including during dose interruptions) with study medications and for 3 months following the last dose of study medication, even if he has undergone a successful vasectomy.

Exclusion Criteria:

1. Prior therapy for pancreatic cancer (e.g., attempted surgery, chemotherapy, radiation therapy).
2. Any contraindication to curative surgery.
3. History of any second malignancy in the last 5 years except in-situ cancer or basal or squamous cell skin cancer. Subjects with history of other malignancies are eligible if they have been continuously disease free for at least 5 years.
4. Severe arterial thromboembolic events (myocardial infarction, unstable angina pectoris, stroke) less than 6 months before study participation.
5. New York Heart Association (NYHA) Class III or IV congestive heart failure, ventricular arrhythmias or uncontrolled blood pressure.
6. Active infection or an unexplained fever >38.5°C during screening visit or on the first scheduled day of dosing in each cycle which, in the Investigator's opinion, might compromise the subject's participation in the trial or affect the study outcome. Subjects with tumor fever may be enrolled at the discretion of the Investigator.
7. Known hypersensitivity to any of the components of nal-IRI, other liposomal products, fluoropyrimidines or leucovorin.
8. Neuropathy > grade 1.
9. Investigational therapy administered within 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is longer, prior to the first scheduled day of dosing in this study.
10. Any other medical or social condition deemed by the Investigator to be likely to interfere with a subject's ability to sign informed consent, cooperate and/or participate in the study in any way, or interfere with the interpretation of the results.
11. Inability or unwillingness to provide written informed consent.
12. Patients who are not appropriate candidates for participation in this clinical study for any other reason as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-17 (Actual); Primary Completion 2021-09-17 (Estimated); Study Completion 2022-09-17 (Estimated)

PRIMARY OUTCOMES:
Treatment safety as assessed by CTCAE v4.03 | An average of 1 year
  Toxicities are evaluated according to CTCAE v4.03

SECONDARY OUTCOMES:
Overall survival | 5 years
  OS is defined as the time between the date of enrollment and the date of death (whatever the cause).
Progression free survival (PFS) | 5 years
  PFS is defined as the time between the date of enrollment and the date of the first radiological and/or pathological progression. Progression is assessed by investigator according to RECIST v1.1 criteria.
Response rate | An average of 1 year
  Response rate will be assessed per RECIST v1.1 criteria and CA19-9 over the entire treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent J Picozzi, MD, Principal Investigator — Virginia mason medical Center
Locations (1):
- Virginia mason medical Center, Seattle, Washington, United States